CLINICAL TRIAL: NCT03331172
Title: Efficacy and Safety of High Intensity Focused Ultrasound (HIFU) Reapplication in Benign Thyroid Nodules That Had Less-than Adequate Shrinkage Following Single-session HIFU Treatment.
Brief Title: HIFU Reapplication in Benign Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 17-234
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Thyroid Nodule
Keywords: HIFU; thyroid nodule; Benign; Reapplication
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Focused Ultrasound (Experimental)
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse — Echopulse is a real-time US-guided High-intensity focused ultrasound (HIFU) system, the HIFU session is a noninvasive procedure that involves application of a focused high-energy ultrasound beam for thermal tissue ablation inside the targeted zone, with minimal effect on the surrounding tissue
  Other Names: High Intensity Focused Ultrasound (HIFU)

SUMMARY:
High Intensity Focused Ultrasound (HIFU) is a new approach in treating benign thyroid nodule without surgery. It is proven effective and safe relative to traditional surgery. From previous HIFU studies, it caused shrinkage of thyroid nodule up to 70% from original size. Unfortunately, 5-10% of nodule do not shrink. Those which do not shrink are usually large in size and therefore a second HIFU treatment may help. This study is going to evaluate the efficacy and safety of reapplication HIFU after the first single HIFU session in 6 months.

The study will be carried out in the following steps:

1. Recruit subject from the clinic according to the study criteria.
2. Arrange the reapplication HIFU treatment within 3 months.
3. Arrange 4 visits after the HIFU treatment in Post 7 days, Post 1 month, Post 3 months, and Post 6 months; Data collection will be in these 4 visits through the questionnaire or interview by research assistant
4. The subjects will have further health management with the same team after the study.

DETAILED DESCRIPTION:
Thyroid nodules are common and although most are benign and remain relatively static in size, some can grow and become large and cause local symptoms over time. In such scenario, thyroidectomy is usually indicated. However, surgery is not only associated with complications but also with high cost and general anesthesia. As a result, there has been a growing interest in exploring less invasive, non-surgical technique for benign thyroid nodules. For solid or predominantly-solid (<30% cystic areas) thyroid nodules, thermal ablation techniques have been shown to be highly effective in causing nodule shrinkage and alleviating symptoms in the long-term. To date, numerous thermal ablation techniques have been described and they include radiofrequency ablation (RFA), percutaneous laser ablation (PLA), microwave ablation and more recently, high intensity focused ultrasound (HIFU). HIFU is now considered the least invasive technique as there is no need for needle insertion into the target lesion during treatment. It works by utilizing focused ultrasound energy to generate heat and induce thermal ablation beneath the skin and other tissue layers. Recent studies (including several from our group) have shown that it is effective in not only inducing significant nodule shrinkage but also in alleviating nodule-related symptoms.

However, despite its overall success, approximately 10 - 15% of solid or predominantly solid nodules do not shrink adequately (i.e. <50% shrinkage from baseline in the first 6-12 months). Although the exact reason why some nodules do not respond remains unclear, it is noted that the majority of these less responsive nodules are larger in size / volume and so, a second or reapplication of ablation might be required to cause further shrinkage and improvement in symptoms [11]. However, the role of HIFU reapplication in nodules with less-than-adequate response (<50% at 6 months) remains undefined. As a result, the present study is aimed to the feasibility and safety of HIFU reapplication in nodules with shrinkage <50% of baseline volume 6 months after single-session HIFU treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients age older than 18 years,
* a nodule that has previously been completely treated by single-session HIFU ablation but has not responded adequately (i.e. <50% volume reduction from baseline after 6 months),
* a benign nodule without signs of malignancy (e.g, nonsuspicious clinical and US appearance, benign results at cytologic examination performed in the last 6 months, normal serum calcitonin level),
* a nodule measuring on US greater than or equal to 10 mm in three orthogonal dimensions,
* less than 30% of the targeted nodule comprising cystic area,
* HIFU accessibility of the targeted nodule (distance between the skin and the anterior surface of the nodule less than 17 mm, with no interference of the collarbone with HIFU unit movements)
* normal thyrotropin concentration and
* absence of vocal cord immobility at laryngoscopy.

Exclusion Criteria:

* head and/or neck disease preventing hyperextension of the neck,
* history of thyroid cancer or other malignant tumors in the neck region,
* history of neck irradiation,
* intranodular macrocalcifications inducing a shadow substantial enough to preclude treatment with HIFU,
* nodules next to the posterior margin of the thyroid lobe with anteroposterior diameter less than 15 mm,
* pregnancy or lactation,
* any contraindication related to intravenous moderate sedation in the first HIFU treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in thyroid nodule volume (mL) | 6 months
  To measure the change in volume (mL) of the index (or treated) thyroid nodule 6 months following HIFU reapplication

SECONDARY OUTCOMES:
The efficacy of reapplication HIFU after the first single session in 6 months | 6 months
  To compare the change in volume (mL) of the treated thyroid nodule between the first single session and the reapplication.
The safety of reapplication HIFU after the first single session in 6 months | 6 months
  To assess the safety of reapplication HIFU by recording any complications after the treatment
The rate of vocal cord palsy in reapplication HIFU after the first single session in 6 months | 6 months
  To examine the rate of vocal cord palsy in reapplication HIFU after the first single session in 6 month
The cosmetic score (in 0-10) of reapplication HIFU after the first single session in 6 months | 6 months
  To evaluate the cosmetic score (in 0-10) of reapplication HIFU after the first single session in 6 months
The pain score (in 0-10) of reapplication HIFU after the first single session in 6 months | 6 months
  To evaluate the pain score (in 0-10) of reapplication HIFU after the first single session in 6 month
The satisfactory (in 0-10) of reapplication HIFU after the first single session in 6 month | 6 months
  The satisfactory level, from scoring in 0-10, to examine how participants' satisfaction in the reapplication HIFU after the first single session in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS (Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] Gharib H, Hegedus L, Pacella CM, Baek JH, Papini E. Clinical review: Nonsurgical, image-guided, minimally invasive therapy for thyroid nodules. J Clin Endocrinol Metab. 2013 Oct;98(10):3949-57. doi: 10.1210/jc.2013-1806. Epub 2013 Aug 16. PMID 23956350
- [Background] Sung JY, Baek JH, Kim KS, Lee D, Yoo H, Kim JK, Park SH. Single-session treatment of benign cystic thyroid nodules with ethanol versus radiofrequency ablation: a prospective randomized study. Radiology. 2013 Oct;269(1):293-300. doi: 10.1148/radiol.13122134. Epub 2013 Apr 24. PMID 23616630
- [Background] Korkusuz H, Sennert M, Fehre N, Happel C, Grunwald F. Local thyroid tissue ablation by high-intensity focused ultrasound: effects on thyroid function and first human feasibility study with hot and cold thyroid nodules. Int J Hyperthermia. 2014 Nov;30(7):480-5. doi: 10.3109/02656736.2014.962626. Epub 2014 Oct 14. PMID 25313977
- [Background] Kovatcheva RD, Vlahov JD, Stoinov JI, Zaletel K. Benign Solid Thyroid Nodules: US-guided High-Intensity Focused Ultrasound Ablation-Initial Clinical Outcomes. Radiology. 2015 Aug;276(2):597-605. doi: 10.1148/radiol.15141492. Epub 2015 Mar 13. PMID 25768327
- [Background] Lang BH, Woo YC, Wong CKH. High-Intensity Focused Ultrasound for Treatment of Symptomatic Benign Thyroid Nodules: A Prospective Study. Radiology. 2017 Sep;284(3):897-906. doi: 10.1148/radiol.2017161640. Epub 2017 Apr 18. PMID 28419814
- [Background] Huh JY, Baek JH, Choi H, Kim JK, Lee JH. Symptomatic benign thyroid nodules: efficacy of additional radiofrequency ablation treatment session--prospective randomized study. Radiology. 2012 Jun;263(3):909-16. doi: 10.1148/radiol.12111300. Epub 2012 Mar 21. PMID 22438360
- [Background] Jeong WK, Baek JH, Rhim H, Kim YS, Kwak MS, Jeong HJ, Lee D. Radiofrequency ablation of benign thyroid nodules: safety and imaging follow-up in 236 patients. Eur Radiol. 2008 Jun;18(6):1244-50. doi: 10.1007/s00330-008-0880-6. Epub 2008 Feb 20. PMID 18286289